CLINICAL TRIAL: NCT04719702
Title: Palliative Sedation Across European Settings: a Prospective Observational Multicentre Study
Brief Title: The Clinical Practice of Palliative Sedation
Acronym: PALLSED
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: European Union (Other); European Association for Palliative Care (EAPC) (Unknown); KU Leuven (Other); University Hospital, Bonn (Other); Clinica Universidad de Navarra, Universidad de Navarra (Other); La Maddalena SPA, Palermo (Unknown)
Responsible Party: Sponsor
Other Study IDs: NL72725.091.20; 825700 (Other Grant/Funding Number: H2020-EU.3.1.3.)
Record Dates: First submitted 2021-01-11; First posted 2021-01-22 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Palliative Sedation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Palliative Sedation (PS) is defined as the intentional lowering of consciousness of a patient in the last phase of life, to relieve patients suffering from refractory symptoms. For those symptoms all possible effective treatments, within an acceptable timeframe, are exhausted.

Several studies have been performed about palliative sedation, mostly focusing on continuous deep sedation, with the use of various measurements to monitor its effect. Efficacy of continuous palliative sedation has been monitored by agitation/distress levels, symptom control, levels of sedation/awareness, comfort, safety and family/caregivers satisfaction. Differences between studies occur, for instance in definition, application and monitoring. Consequently reported outcomes and associated treatment goals differ between studies which makes it difficult to compare the results.

Within this international multicenter observational study, the investigators aim to evaluate the effects of palliative sedation on patient's comfort levels. Participants with different forms and intensity of palliative sedation (intermittent and continuous, from light to deep) are included in a prospective design as part of an international study.

Objectives:

1. To evaluate the effect of palliative sedation on participants' comfort and other symptoms in different international hospices, palliative care units and hospital ward settings.
2. To assess the clinical practice of palliative sedation in different international care settings and the accompanying costs and consequences.

Study design: Prospective observational multicentre study in hospices, palliative care units and hospital ward settings in five European countries (Belgium, Germany, Italy, Spain, The Netherlands).

ELIGIBILITY:
Phase 1: Participants are eligible for participation in this study when they meet all the following criteria:

* Adults;
* with advanced cancer;
* and a limited life expectancy (1- 2 months);
* according the health care team, intractable distress caused by one or more refractory symptoms can be expected or is present during the hospitalization.

Participants can enter Phase 2 of this study when fulfilling the following preconditions:

* inclusion criteria for phase 1 are met and informed consent is given by the participant;
* participant is suffering from intractable distress caused by one or more refractory symptoms according the health care team and/or participant and relatives;
* sedative medication is started with the aim to relieve burden of otherwise intractable suffering (palliative sedation)

Exclusion Criteria:

* a potential participant is unable to give informed consent;
* a potential participant is unable to speak and read in the native language of the participating country.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutively admitted patients to one of the participating palliative care settings (PC units / consulted by PC team at the hospital wards / Hospices) will be screened for eligibility. Preferably, eligible particpants and/or their relatives are informed about the study in an early stage of their palliative care trajectory. Therefore, we use two phases: phase 1: admitted patients with advanced cancer and limited life expectancy; phase 2: deteriorating patient's and the decisionprocess about palliative sedation is started.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Levels of discomfort | T0: Baseline before start PS (max. 8 hours before); T1: First measurement after start PS, within 6 hours after start PS; T2-T..: Measurements are continued twice a day during PS until the date of death, on average less than 1 week
  Change in discomfort levels of participants receiving a form of palliative sedation (PS) will be measured by the Discomfort Scale-Dementia of Alzheimer Type (DS-DAT). The tool covers nine categories: noisy breathing, negative vocalizations, content facial expression, sad facial expression, frightened facial expression, frown, relaxed body language, tense body language, and fidgeting. Items are scored by indicating behaviors that are present/absent with a resulting range of scores from 0 to 27. Higher scores represent higher amount of discomfort.

SECONDARY OUTCOMES:
Levels of agitation and sedation | T0: Baseline before start PS (max. 8 hours before); T1: First measurement after start PS, within 6 hours after start PS; T2-T..: Measurements are continued twice a day during PS until the date of death, on average less than 1 week
  Change in levels of agitation and sedation of participants receiving a form of palliative sedation will be measured by the Richmond Agitation Sedation Scale-modified version for Palliative Care (RASS-PAL). This scale is a modified version of the RASS. The RASS-PAL is a 10-point scale ranging from -5 to +4. Levels -1 to -5 denote 5 levels of sedation, starting with "awakens to voice" and ending with "unarousable." Levels +1 to +4 describe increasing levels of agitation. The lowest level of agitation starts with apprehension and anxiety, and peaks at combative and violent. RASS-PAL level 0 is "alert and calm."

OTHER OUTCOMES:
Changes in dosage of administered sedative medication during Palliative Sedation | Daily Registration from start PS until the date of death, on average less than 1 week
  When PS is started a list of medications is completed daily. Part of this medication list contains information about changes in dosages of sedative medication. Medication dosage can be increased or decreased. The changed dosage is registered in numbers; units (mg or mg/hr); and date and time of the change.
Changes in sort of administered sedative medication during Palliative Sedation | Daily Registration from start PS until the date of death, on average less than 1 week
  When PS is started a list of medications is completed daily. Part of this medication list contains information about changes in sort of sedative medication used for palliative sedation. The sort medication dosage can be changed by starting a new sort of medication or stopping a sort of administered sedative medication. Changes in the sort of sedative medication are registered with the medication name and the date and time of change.
Changes in route of administered medication during Palliative Sedation | Daily Registration from start PS until the date of death, on average less than 1 week
  When PS is started a list of medications is completed daily. Part of this medication list contains information about changes in route of the administered medication used for palliative sedation. The route of administered medication can be changed from subcutaneous to intravenous or vice versa; from bolus to continuous. Changes in the route of sedative medication are registered with the route and the date and time of change.
Amount of staff time (in minutes) needed for tasks in different phases of PS | T1: During the decision process; T2: Start/Initiation of PS; T3-T..: Daily registration of time until the death date, on average 1 week
  During the different phases of PS (decision making; initiating; monitoring; aftercare) the attending HCPs registrate their individual spent time needed for tasks within the process.
Satisfaction with care during the palliative sedation period by one of the relatives | T1: Once, One month after the participant's death the relative receives the questionnaire.
  The Satisfaction of Family Caregivers (FAMCARE-2) Scale is a tool used to measure family satisfaction with advanced cancer care. The FAMCARE-2 measures the degree to which family members are content with the palliative care team behaviors directed toward the patient and themselves. Items are referring to four different areas of care such as availability of care, physical patient care, psychosocial care and information giving. Items are scored at a five-point Likert-scale with the following responses: very satisfied, satisfied, undecided, dissatisfied and very dissatisfied. A total score ranging from 17 to 85 and scores for the four subscales can be calculated. Higher sum scores indicate higher satisfaction.
Evaluation of the palliative sedation period of the patient by one of the Health Care Professionals (HCP) | T1: Once, within one week after the participant's death the HCP receives the questionnaire.
  One of the attending HCPs, which was present during the start of the palliative sedation, is asked to complete an ad hoc questionnaire about the palliative sedation in the specific participant's case. The items that are asked to score on a Likert scale are: 1. Agreement with the decision (strongly disagree - disagree - undecided - agree - strongly agree); 2. The overall achieved effect of palliative sedation at patient's comfort levels (excellent - good - fair - poor - very poor); 3. The quality of dying (excellent - good - fair - poor - very poor).

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen GJ Hasselaar, MSc, PhD, Principal Investigator — Radboud University Medical Center
Locations (8):
- Katholieke Universiteit Leuven, Leuven, Belgium
- Universitätsklinikum Bonn, Bonn, Germany
- La Maddalena Spa, Palermo, Italy
- Netherlands (4):
  - Rijnstate Ziekenhuis, Arnhem
  - Radboud University Medical Centre, Nijmegen
  - Hospice Bethlehem - Kalorama, Nijmegen
  - Hospice de Hazelaar, Liemerije, Zevenaar
- Clinica Universidad de Navarra, Pamplona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rijpstra M, Vissers K, Belar A, Van der Elst M, Surges SM, Adile C, Roji R, Grassi Y, Bronkhorst E, Mercadante S, Radbruch L, Menten J, Centeno C, Kuip E, Hasselaar J. Assessment of the efficacy of palliative sedation in advanced cancer patients by evaluating discomfort levels: a prospective, international, multicenter observational study. BMC Med. 2024 Dec 31;22(1):608. doi: 10.1186/s12916-024-03829-7. PMID 39741317
- [Derived] Rijpstra M, Vissers K, Centeno C, Menten J, Radbruch L, Mercadante S, Van der Elst M, Adile C, Arantzamendi M, Kuip E, Payne S, Preston N, Hasselaar J. Monitoring the clinical practice of palliative sedation (PALSED) in patients with advanced cancer: an international, multicentre, non-experimental prospective observational study protocol. BMC Palliat Care. 2023 Jan 28;22(1):8. doi: 10.1186/s12904-022-01125-w. PMID 36709271